CLINICAL TRIAL: NCT03544957
Title: Evaluation of the Triage Risk Screening Tool (TRST) as Screening Instrument Elderly Subject Fragility at the Accident and Emergency Department
Brief Title: Evaluation of the Triage Risk Screening Tool
Acronym: TRST-U
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-02Obs-CHRMT
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2018-04

CONDITIONS: Elderly Subject Fragility
Keywords: Screening instrument

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study tried to describe diagnostic properties of TRST completed by an emergency doctor, for screening process for fragility of elderly subjects admitted at the accident and emergency department.

DETAILED DESCRIPTION:
A constant increase of emergencies admission of elderly subjects is registered. The current problem is the identification and early screening of these patients upon admission at the accident and emergency department for early tracking in geriatric network. This early assessment could allow a shorter waiting time, a better orientation of patients and a decrease in the number of re-hospitalization.

There are many screening process for fragility tests but there seem to be nonspecifically. The advantage of TRST is its simplicity and speed of filling.

In 2015, Duc et al. have found that TRST may be a screening instrument for elderly subject and is going to require geriatric mobile team (GMT) for evaluation. Unfortunately, the threshold may be too sensitive and GMT solicitation is too high.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are more than 75 years old
* Admitted to the emergency department for medical or surgical reason
* Admitted from Monday to Friday (8h30 AM- 6h PM)

Exclusion Criteria:

* Patient with specific care (vital emergency, urgent surgery)
* Patient or his support person opposing the use of data

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly subject admitted to the emergency department
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
TRST-U | Day 1
  Triage Risk Screening Tool completed by an emergency doctor

SECONDARY OUTCOMES:
TRST-G | Day 1
  Triage Risk Screening Tool completed by a geriatrician
SEGA instrument | Day 1
  Evaluation of TRST versus SEGA instrument (gold standard)

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Metz Thionville, Metz, Moselle, France

IPD SHARING:
Plan to Share IPD: No